CLINICAL TRIAL: NCT04991714
Title: Einfluss Der Süßintensität Einer Saccharose-Lösung Auf Die Blutglukoseregulation Und Energieaufnahme in Gesunden Männern
Brief Title: Effect of Sweetness Intensity of a Sucrose Solution on Blood Glucose Regulation and Energy Intake
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Lieder, Deptuy Head Department of Physiological Chemistry, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 706014-1
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Blood Glucose, Low; Hunger
MeSH Terms: interventions — lactisole; rebaudioside M; Sucrose; Dietary Sucrose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sucrose (Experimental): 10% solution in water
  Interventions: Other: Sucrose
- Sucrose + Reb M (Experimental): 10% sucrose + 60 mg/L Rebaudioside M
  Interventions: Drug: Rebaudioside M; Other: Sucrose
- Sucrose + Lactisole (Experimental): 10% sucrose + 30 mg/ L Lactisole
  Interventions: Drug: Lactisole; Other: Sucrose
- Sucrose + Reb M + Lactisole (Experimental): 10% sucrose + 60 mg/L Rebaudioside M + 30 mg/ L Lactisole
  Interventions: Drug: Lactisole; Drug: Rebaudioside M; Other: Sucrose

INTERVENTIONS:
Drug: Lactisole — sweet taste inhibitor (decreases sweetness)
  Other Names: 2-(4-methoxyphenoxy)propionic acid; CAS Number: 150436-68-3
  Arms: Sucrose + Lactisole; Sucrose + Reb M + Lactisole
Drug: Rebaudioside M — Sweetener (increases sweetness)
  Other Names: CAS Number: 1220616-44-3
  Arms: Sucrose + Reb M; Sucrose + Reb M + Lactisole
Other: Sucrose — 10% Sucrose corresponding to a regular soft drink
  Other Names: table sugar

SUMMARY:
The aim of the present study is to investigate the influence of the modulation of the sweetness intensity of a carbohydrate (sucrose)-containing solution on metabolic effects, in particular the regulation of blood glucose concentration and regulation of hunger & satiety.

DETAILED DESCRIPTION:
The study is designed as a randomised cross-over intervention study with four interventions. The study investigates the influence of sweetness modulation by Rebaudioside M (sweetness enhancement) and Lactisol (sweetness inhibition) of a 10% sucrose solution, corresponding to the concentration of a regular soft drink, on blood glucose regulation (blood glucose concentration and regulating hormones) in healthy male volunteers. Furthermore, the study assesses ad libitum energy intake, individual feelings of hunger and satiety, metabolic responses to the interventions, and preference for sweet-tasting foods such as sugar and sweeteners. In addition, the participants' individual thresholds for sweet taste, as well as morphological markers for taste sensitivity and body composition will be recorded as potential influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* non-smoking
* normal taste responses towards sweet taste

Exclusion Criteria:

* female
* regular smokers
* disturbed glucose and/or lipid metabolism
* regular intake of medication
* known allergies against one of the test compounds
* ageusia
* alcohol or drug addiction
* intake of antibiotics within the past 2 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentration | over a time span of 120 minutes after drinking the test solution
  Glucose concentration [mg/dL] in plasma samples before, and 15, 30, 60, 90, and 120 minutes after drinking the test solution
Insulin concentration | over a time span of 120 minutes after drinking the test solution
  Insulin concentration [mmol/L] in plasma samples before, and 15, 30, 60, 90, and 120 minutes after drinking the test solution
GLP-1 concentration | over a time span of 120 minutes after drinking the test solution
  Glucagon-like peptide 1 concentration in plasma samples [mmol/L] before, and 15, 30, 60, 90, and 120 minutes after drinking the test solution
GIP-concentration | over a time span of 120 minutes after drinking the test solution
  Gastric inhibitory polypeptide concentration in plasma samples [mmol/L] before, and 15, 30, 60, 90, and 120 minutes after drinking the test solution

SECONDARY OUTCOMES:
Food intake | 120 minutes after drinking of the test solution
  Ad libitum Food intake from a standardized breakfast
Metabolic changes | over a time span of 120 minutes after drinking the test solution
  Metabolome analysis in plasma samples [mmol/L] before, and 15, 30, 60, 90, and 120 minutes after drinking the test solution

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lieder, PhD, Principal Investigator — University of Vienna
Locations (1):
- Christian Doppler Laboratory for Taste Research, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No